



# PROTOCOL OF A THESIS FOR PARTIAL FULFILMENT OF MD DEGREE IN INTERNAL MEDICINE

**Title of the Protocol:** Effect of Tight Glycemic Control on Microvascular Complications in Type 2 Diabetes Mellitus: A Randomized Controlled Trial in an

**Egyptian Cohort** 

**Date of document:** May 1st, 2022

Postgraduate Student: Ola Mohamed Mostafa Shaheen

**Degree:** Master of internal medicine- Faculty of Medicine – Ain Shams University

**DIRECTOR: Dr. Manal Mohamed Abu Shady** 

**Academic Position:** Professor

**Department:** Internal Medicine, Endocrinology Department – Ain Shams University

Co-DIRECTOR: Dr. Mona Mohamed Abdelsalam

**Academic Position:** Professor

**Department:** Internal Medicine, Endocrinology Department – Ain Shams University

**Co-DIRECTOR: Dr. Meram Mohamed Bekhet** 

**Academic Position:** Assistant Professor

**Department:** Internal Medicine, Endocrinology Department – Ain Shams University

Co-DIRECTOR: Dr. Salah Hussein Elhalawany

**Academic Position: Lecturer** 

**Department:** Internal Medicine, Endocrinology Department – Ain Shams University

Co-DIRECTOR: Dr. Hany Khairy Mansour

**Academic Position: Lecturer** 

**Department:** Internal Medicine, Endocrinology Department – Ain Shams University

Faculty of Medicine Ain Shams University 2021





# What is already known on this subject? AND

## What does this study add?

Near normalization of blood glucose levels has been known to reduce the long-term risk of diabetic retinopathy. However, transient worsening of preexisting retinopathy has also been demonstrated when glucose control is intensified (**Bethel A. et al., 2021**).

The pathophysiology of this phenomenon is not well understood. Furthermore, the circumstances under which it appears remain to be not fully elucidated. Since its discovery, early worsening has been described in patients with type 1 and type 2 diabetes, including those undergoing various diabetic therapies, those who have undergone bariatric surgery, and pregnant women (**Feldman-Billard** *et al.*, **2018**).

Hence, this study will assessthe relationship between the glycemic control in patients with diabetes mellitus and the contemporary statements on the value of tight glycemic control, when compared with less tight control with regard to microvascular outcomes including diabetic retinopathy, nephropathy and neuropathy.

## 1.INTRODUCTION/ REVIEW

Diabetes mellitus (DM) is a metabolic disorder characterized by chronic hyperglycemia due to either insulin deficiency or resistance or both (Goyal&Jialal 2021). Hyperglycemia induces tissue damage through mitochondrial superoxide production, affecting retina, glomerulus, and neurons. It requires continuing medical care and ongoing self-care management to prevent and delay acute and long-term micro and macrovascular complications (Fasil A et al., 2019).

Chronic diabetes complications like retinopathy, nephropathy, neuropathy, self-reported chest pain, vision decrement, painful paresthesia, and psychiatric





events result in decrement of health-related quality of life (Jacobson et al., 2013).

Diabetic retinopathy (DR) is the most common microvascular complication of DM and is a leading cause of blindness in the working age population worldwide (Leasheret al., 2016). It is a progressive sight-threatening eye disease caused by hyperglycemia, which damages the retinal microvasculature leading to vascular permeability, retinal ischemia, neovascularization, retinal detachment, and blindness (Augustine et al., 2020).

After the DCCT (Diabetes Control and Complications Trial) found that tight glycemic control (a glycohemoglobin A1c (HbA1c) <7%) could prevent or slow the progression of nephropathy, retinopathy, and neuropathy in patients with diabetes mellitus, a consensus, extended to patients with type 1 and type 2 diabetes mellitus, emerged: normalizing glycemia prevents diabetes mellitus complications (**Garber** *et al.*, 2013). Guidelines, quality improvement interventions, quality-of-care measures and patient-directed marketing have since focused on achieving tight glycemic control. (**Rodriguez &Montori2016**).

Appropriate glycemic control and management is fundamental to prevent and delay DM complications. Poor glycemic control is highly correlated with high burden of diabetes complications. However, data are scanty regarding factors for poor glycemic control and the relationship between glycemic control and DM complications (Fasil A et al., 2019).

#### 2.AIM / OBJECTIVES

This randomized controlled study will examine the relation between tight glycemic control and microvascular complications of Diabetes in comparison with patients with good (less tight) glycemic control.

**Research question**: Does tight glycemic control worsens microvascular complications of Diabetes?





## **3.METHODOLOGY:**

## Patients and Methods/ Subjects and Methods/ Material and Methods

## • Type of Study:

Randomized controlled trial.

## • Study Setting:

The study will be conducted at Ain Shams University Hospitals "outpatient diabetes clinic and inpatient department."

# Study duration:

This study will be conducted during the period from May 2022 to October 2023

• Labs (see later), thorough clinical examination with special emphasis on microvascular complications (neurological and Fundus examination) will be done for every patient at time of recruitment and 6 months following glycemic control.

# • Study Population:

- 80subjects with uncontrolled Diabetes Mellitus with HbA1c 8% or above all will receive standard medical care (nutritional therapy and pharmacological therapy) and will be divided into two groups:
  - (a) Group (A) will undergo tight glycemic control (HbA1c <7%) done by nutritional education and medication adjustment.
  - (b) Group (B) will undergo conventional glycemic control (HbA1c <7.5 %).





Subjects will be collected from patients with Diabetes Mellitus referred to Ain Shams University Hospitals for evaluation with the following criteria:

## • Inclusion criteria:

- **1.** Both sexes.
- **2.** Age 18-60 years old.
- **3.** Patients diagnosed with Diabetes Mellitus (Type 2) according to ADA guidelines.
- **4.** Patients willing to participate after signing a written consent to be enrolled in the study after being explained to them in an interview.
- **5.** Diabetic patients with mild and moderate non proliferative diabetic retinopathy

#### **Exclusion criteria:**

- 1. Patients with age above 60 or below 18 years old.
- **2.** Patients with severe non proliferative diabetic retinopathy up to advanced proliferative diabetic retinopathy.
- **3.** Patients diagnosed with type 1 DM.
- **4.** Patients with malignant tumors.
- **5.** Patients with end stage renal disease and end stage liver disease.
- **6.** Patients with history of myocardial infarction.
- **7.** Patients with recurrent attacks of hypoglycemia and hypoglycemia unawareness.





# **Sampling Method:**

Purposive sampling

## **Sample Size:**

The study will be conducted on 80 subjects.

# **Ethical and Safety Consideration:**

This study will be done after approval of the Ethical Committee of the Department of Internal Medicine, Faculty of Medicine, Ain Shams University. Informed consent will be taken from all participants before recruitment in the study, and after explaining the purpose and procedures of the study. The investigator will retain the original signed informed consent form. All data will be collected confidentially. The study will be based on the investigator self-funding.

# **Study procedures and interventions:**

- **1.** After approval of study protocol, patients will be enrolled into the study according to inclusion and exclusion criteria.
- **2.** All participants will sign written informed consent that is approved by the local ethics committee.
- **3.** All patients will be subjected to:
  - > Detailed history taking of the patient medical condition.
  - ➤ Anthropometric and blood pressure measurements:
    - ✓ Weight and height of all patients will be measured using a calibrated scale. Body mass index (BMI) will be calculated by dividing weight in kilograms by height in meters squared.





- ✓ Blood pressure will be measured in both standing and seated position after a 5-min rest using an aneroid sphygmomanometer and stethoscope.
- ✓ Basal heart rate measurement

# **>** Biochemical assays:

- ✓ Laboratory measurements will include:
  - ❖ Fasting, 2 hour post prandial glucose levels and HbA1C.
  - \* Kidney function tests including serum urea and creatinine.
  - ❖ Albumin/creatinine ratio.
  - ❖ Estimated GFR calculation using MDRD 4 variable equation.
  - Complete blood count.
- > Fundus examination using Optomed aurora portable fundoscopy.
- > Neurological assessment using DN4 (Douleur Neuropathique 4 questions).
- Labs, neurological and Fundus examination will be done at time of recruitment and 6 months following glycemic control.
- Outcomes:

Effect of tight glycemic control on microvascular complications of Diabetes.

Statistical analysis:





To summarize characteristics of study patients based on TyG quartiles, one-way analysis of variance (ANOVA) and chi-square (c2) tests will be used, where appropriate. To determine the association of liver fibrosis with TyG, multivariable-adjusted odds ratios (ORs) will be applied. Two-sided significance at P < 0.05 will be significant.

## **Statistical Package:**

Data will be analyzed with the use of IBM SPSS Statistics.

## **4.REFERENCES:**

- Bain S,Klufas M, Allen H, et al. (2019): Worsening of diabetic retinopathy with rapid improvement in systemic glucose control: Diabetes ObesMetab.; 21(3): 454–466.
- Bethel A, Diaz R, Lakshmanan M, et al. (2021): HbA<sub>1c</sub> Change and Diabetic Retinopathy During GLP-1 Receptor Agonist Cardiovascular Outcome Trials: A Meta-analysis and Meta-regression. Diabetes care. ;44(1): 290-296.
- Fasil A, Biadgo B and Abebe M. (2019): Glycemic control and diabetes complications among diabetes mellitus patients attending at University of Gondar Hospital, Northwest Ethiopia. Diabetes, Metabolic Syndrome and Obesity: Targets and Therapy, Volume 12: pages 75-83.
- Feldman-Billard S, Larger É and Massin P. (2018): Early worsening of diabetic retinopathy after rapid improvement of blood glucose control in patients with diabetes. *Diabetes Metab*.;44:4-14.
- Garber AJ, Abrahamson MJ, Barzilay JI, et al. (2013): comprehensive diabetes management algorithm. EndocrPract.; 19:327–336.
- GoyalR and Jialal I. (2021) Diabetes Mellitus Type 2. Stat pearls.





- Jacobson AM, Braffett BH, Cleary PA, et al. (2013): DCCT/EDIC Research Group. The long-term effects of type 1 diabetes treatment and complications on health-related quality of life. *Diabetes Care*.;36(10):3131–3138.
- Rodriguez-Gutierrez R and Montori M. (2016): Glycemic Control for Patients with Type 2 Diabetes: Our Evolving Faith in the Face of Evidence. CircCardiovascQual Outcomes.; 9(5): 504–512.
- Leasher JL, Bourne RRA, Flaxman SR, et al. ((2016): Global estimates on the number of people blind or visually impaired by diabetic retinopathy: A meta-analysis from 1990 to 2010. Diabetes Care 39:1643–9.
- Augustine J, Troendle E, Curtis T etal. (2020): The Role of Lipoxidation in the Pathogenesis of Diabetic Retinopathy. Front Endocrinology (Lausanne),11:621938.